CLINICAL TRIAL: NCT03885479
Title: Impact of Different Dietary IgGs on the Pathogenesis of Inflammatory Bowel Disease
Brief Title: Impact of Different Dietary IgGs on the Pathogenesis of IBD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hebatallah Mohammed Abdelwahab Mohammed Abdelrahman, Principal investigator, Assiut University
Other Study IDs: IBDIgG
Record Dates: First submitted 2019-03-18; First posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Inflammatory Bowel Diseases; Food Intolerance
Keywords: Inflammatory bowel disease; Food specific IgGs
MeSH Terms: conditions — Inflammatory Bowel Diseases; Food Intolerance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IBD patients: 1. Full history taking and examination
  2. Colonoscopy, biopsy and histopathology to determine the extent of the lesion
  3. An enzyme-linked immunosorbent assay (ELISA) for the semi-quantitative analysis of serum food-specific IgGs against 7 food-derived antigens (Wheat, rice, beans, cow milk, eggs, chicken and beef)
  4. Patients will be categorized into 3 groups (UC patients, Crohn disease patients and controls)
  5. All of the following factors will be taken into consideration; type and duration of the treatment, age of diagnosis, BMI, smoking status and activity of the disease at the time of the study
  Interventions: Diagnostic Test: ELISA for the semi-quantitative analysis of serum food-specific IgGs against food-derived antigens
- Controls: An enzyme-linked immunosorbent assay (ELISA) for the semi-quantitative analysis of serum food-specific IgGs against 7 food-derived antigens (Wheat, rice, beans, cow milk, eggs, chicken and beef)
  Interventions: Diagnostic Test: ELISA for the semi-quantitative analysis of serum food-specific IgGs against food-derived antigens

INTERVENTIONS:
Diagnostic Test: ELISA for the semi-quantitative analysis of serum food-specific IgGs against food-derived antigens — An enzyme-linked immunosorbent assay (ELISA) for the semi-quantitative analysis of serum food-specific IgGs against 7 food-derived antigens (Wheat, rice, beans, cow milk, eggs, chicken and beef)

SUMMARY:
Identify the association between certain food IgGs (Wheat, rice, broad beans, cow milk, eggs, chicken and beef) and the immunological response in patients with IBD

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is comprised of two major disorders: ulcerative colitis and Crohn disease. Ulcerative colitis and Crohn disease have distinct pathologic and clinical characteristics but their pathogenesis remains poorly understood.

In 2015, an estimated 1.3% of US adults (3 million) reported being diagnosed with IBD (either Crohn's disease or ulcerative colitis). This was a large increase from 1999 (0.9% or 2 million adults).The incidence and prevalence of Crohn disease and ulcerative colitis (UC) appear to be lower in Asia and the Middle East , however, in some newly industrialized countries in Africa, Asia, and South America, the incidence of IBD has been rising.

Ulcerative colitis is a chronic inflammatory condition characterized by relapsing and remitting episodes of inflammation limited to the mucosal layer of the colon. It almost invariably involves the rectum and typically extends in a proximal and continuous fashion to involve other portions of the colon.

Crohn disease is characterized by transmural inflammation and by skip lesions. The transmural inflammatory nature of Crohn disease may lead to fibrosis and strictures, and to obstructive clinical presentations that are not typically seen in ulcerative colitis. The transmural inflammation more commonly results in sinus tracts, giving rise to microperforations and fistulae.

Food antigens are thought to trigger an immunologic response resulting in the development of IBD. However, specific pathogenic antigens have not been identified. While studies attempting to associate specific diets with the development of IBD have had inconsistent results, the data suggest that a "Western" style diet (processed, fried, and sugary foods) is associated with an increased risk of developing Crohn disease, and possibly ulcerative colitis.

To date, studies concerning food intolerance in IBD have largely focused on classic food allergies based on IgE mediated antibody responses. The levels of total or food-specific IgEs have been observed to be increased in the sera of IBD patients, and IgE-mediated food allergies are more frequent in IBD patients than in those without IBDs. Nevertheless, reactions mediated by food specific IgGs, featuring a more delayed response following exposure to a particular antigen, are also expected to contribute to adverse reactions in IBD, and food-specific IgGs help physicians identify the candidate food for elimination in IBD patients. Furthermore, IgG-mediated adverse reactions have also been reported to be involved in some cases of food hypersensitivity.

Elimination diet can help in the remission of the disease. An elimination diet involves removing a food from the diet for a period of time and seeing whether symptoms resolve during that time. In patients receiving enteral nutrition, it involves introducing one new food at a time to identify foods that precipitate IBD symptoms. Many patients can identify foods that they believe may precipitate or worsen their disease and it is reasonable for them to avoid such foods. Using an elimination diet to identify at-risk foods may decrease the possibility of a "flare" of IBD.

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory bowel disease patients (Ulcerative colitis and Crohn's disease)
* Patients aged ≥ 18 years old

Exclusion Criteria:

• Patients who started TNF-α inhibitor (Infliximab)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Case group: IBD patients Control group: Normal individuals
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Level of serum food specific IgGs in patients with IBD | baseline
  Level of serum food specific IgGs in patients with Inflammatory bowel diseasea against 7 food-derived antigens (Wheat, rice, beans, cow milk, eggs, chicken and beef)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Elyamany, Professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Silverberg MS, Satsangi J, Ahmad T, Arnott ID, Bernstein CN, Brant SR, Caprilli R, Colombel JF, Gasche C, Geboes K, Jewell DP, Karban A, Loftus EV Jr, Pena AS, Riddell RH, Sachar DB, Schreiber S, Steinhart AH, Targan SR, Vermeire S, Warren BF. Toward an integrated clinical, molecular and serological classification of inflammatory bowel disease: report of a Working Party of the 2005 Montreal World Congress of Gastroenterology. Can J Gastroenterol. 2005 Sep;19 Suppl A:5A-36A. doi: 10.1155/2005/269076. PMID 16151544
- [Background] Dahlhamer JM, Zammitti EP, Ward BW, Wheaton AG, Croft JB. Prevalence of Inflammatory Bowel Disease Among Adults Aged >/=18 Years - United States, 2015. MMWR Morb Mortal Wkly Rep. 2016 Oct 28;65(42):1166-1169. doi: 10.15585/mmwr.mm6542a3. PMID 27787492
- [Background] Nguyen GC, Chong CA, Chong RY. National estimates of the burden of inflammatory bowel disease among racial and ethnic groups in the United States. J Crohns Colitis. 2014 Apr;8(4):288-95. doi: 10.1016/j.crohns.2013.09.001. Epub 2013 Sep 24. PMID 24074875
- [Background] Ananthakrishnan AN, Khalili H, Konijeti GG, Higuchi LM, de Silva P, Korzenik JR, Fuchs CS, Willett WC, Richter JM, Chan AT. A prospective study of long-term intake of dietary fiber and risk of Crohn's disease and ulcerative colitis. Gastroenterology. 2013 Nov;145(5):970-7. doi: 10.1053/j.gastro.2013.07.050. Epub 2013 Aug 2. PMID 23912083
- [Background] Mekkel G, Barta Z, Ress Z, Gyimesi E, Sipka S, Zeher M. [Increased IgE-type antibody response to food allergens in irritable bowel syndrome and inflammatory bowel diseases]. Orv Hetil. 2005 Apr 24;146(17):797-802. Hungarian. PMID 17918636
- [Background] Bentz S, Hausmann M, Piberger H, Kellermeier S, Paul S, Held L, Falk W, Obermeier F, Fried M, Scholmerich J, Rogler G. Clinical relevance of IgG antibodies against food antigens in Crohn's disease: a double-blind cross-over diet intervention study. Digestion. 2010;81(4):252-64. doi: 10.1159/000264649. Epub 2010 Jan 30. PMID 20130407
- [Background] Koretz RL, Avenell A, Lipman TO, Braunschweig CL, Milne AC. Does enteral nutrition affect clinical outcome? A systematic review of the randomized trials. Am J Gastroenterol. 2007 Feb;102(2):412-29; quiz 468. doi: 10.1111/j.1572-0241.2006.01024.x. PMID 17311654